CLINICAL TRIAL: NCT03231826
Title: Exploring Arrhythmias After Hospital Discharge in Post-Myocardial Infarction Patients - the MADDEC Project
Brief Title: Arrhythmias in Post-Myocardial Infarction Patients
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: Tays Heart Hospital (Unknown); GE Healthcare Finland Ltd (Unknown); Fimlab Ltd (Unknown); VTT Technical Research Centre of Finland (Other); Bittium Ltd (Unknown); Tekes - Finnish Funding Agency for Innovation (Unknown); Politecnico Milano (Unknown)
Responsible Party: Principal Investigator, Jussi Hernesniemi, Professor, Tampere University
Other Study IDs: R17023
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Infarction; Coronary Artery Disease; Arrythmia; ECG Electrical Alternans; Atrioventricular Block; Atrial Fibrillation; Atrial Flutter; Ventricular Tachycardia; Ventricular Fibrillation; Ventricular Arrythmia
Keywords: Home monitoring; ECG; Myocardial Infarction; Arrythmia
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Arrhythmias, Cardiac; Atrioventricular Block; Atrial Fibrillation; Atrial Flutter; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Recording of continuous ECG-signals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients are screened for significant arrhythmias and other possibly significant ECG-patterns directly after discharge and two weeks after myocardial infarction using wearable devices. The home monitoring data will be linked with extensive data from electronic health records collected before, during hospital stay and after discharge.

The purpose of the study is to clarify whether home monitoring of continuous ECG-signals can be used to predict and prevent serious adverse events after myocardial infarction.

DETAILED DESCRIPTION:
Patients with acute myocardial infarction have exceptionally high mortality rates exceeding 10% during the first year post-MI. The incidence of sudden cardiac death after acute myocardial infarction is the same with ST-elevation and non-ST elevation myocardial infarction. The risk of disabling stroke and sudden cardiac death is high especially during the first months after myocardial infarction. Preventing these outcomes is of high priority, considering the fact that the quality of life can remain high in these patients, if serious adverse events can be avoided.

The high mortality and comorbidity rates among cardiac patients provide an opportunistic environment for testing the utility of of home monitoring by mobile devices, data integration and resulting mass data. Long follow-up times are not required, which facilitates the linking of potential risk factors with outcome.

The prospective part of the MADDEC (MAss Data in Detection and prevention of serious adverse Events in Cardiovascular disease) project aims at exploring mechanism of sudden death in the first month after a myocardial infarction and at detecting arrhythmias heralding life-threatening arrhythmias. Additionally, the project will define the incidence of new atrial fibrillation post myocardial infarction. The main outcomes of the study are all cause mortality, cardiovascular mortality, rehospitalization due to any or cardiovascular causes.

Prospective home monitoring of patients after ST-elevation or non-ST elevation myocardial infarction will commence in May 2017 and continue until the end of 2019. For arrhythmia detection, two different methods will be used: 12-channel Holter recording (GE Seer 12®, GE Healthcare Finland) and the eMotion Faros® device (Bittium Biosignals Ltd/Mega Elec-troncs Ltd, Finland). The aim is to record continuous 12-channel Holter data from 200-250 patients with ST-elevation myo-cardial infarction and 1-3 channel ECG signal data with the mobile Faros 360 device from 550-600 patients with any type of myocardial infarction. Exclusion criteria are short life expectancy, unwillingness to participate and need for permanent insti-tutional care. The first 24-48 hour recording will commence at hospital discharge or transferral to another health care unit. The second recording will take place two weeks after the index event. As a part of the protocol, the subjects will also perform simple tests measuring their functional status and possible disability at study enrollment. All accrued ECG-data will be inte-grated into a research database for further analysis, linking it with outcome data. The Faros 360 mobile device will also ena-ble recording patient activity, such as movement and respiratory rate, simultaneously using an accelerometer.

ELIGIBILITY:
Inclusion Criteria: Patients treated for myocardial infarction (NSTEMI and STEMI)

Exclusion Criteria: Short life expectancy, unwillingness to participate and need for permanent institutional care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated at the study center (Tays Heart Hospital) between June 2017 and June 2019 fulfilling the eligibility criteria are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | One month and one year and five after myocardial infarction
  Mortality due to heart failure, complication of myocardial infarction, recurrent myocardial infarction, stroke or probable cardiac arrhythmia

SECONDARY OUTCOMES:
Incident asymptomatic atrial fibrillation | Within two weeks after myocardial infarction
  Incidence of new-onset atrial fibrillation
Incident ventricular arrhythmias | Within two weeks after myocardial infarction
  Ventricular tachycardias (NSVT and longer), ventricular fibrillation and Ventricular extrasystoles.
Incident bradyarrhytmias | Within two weeks after myocardial infarction
  New bradyarrhytmias including AV block and sinus arrests.
Rehospitalization | One month and one year and five after myocardial infarction
  Rehospitalization due to any cause
Rehospitalization (CVD) | One month and one year and five after myocardial infarction
  Rehospitalization due cardiovascular cause
Incidence of symptomatic atrial arrhythmias | One month and one year and five after myocardial infarction
  Atrial fibrillation, atrial flutter and other atrial arrhythmias leading to patient seeking medical attention and treatment
Incidence of symptomatic ventricular arrhythmias | One month and one year and five after myocardial infarction
  Ventricular fibrillation, ventricular tachycardias and other ventricular arrhythmias medical
Overall mortality | One month and one year and five after myocardial infarction
  Mortality due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jussi A Hernesniemi, MD PhD, Principal Investigator — Tays Heart Hospital and Tampere University
Locations (1):
- Tays Heart Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided
The use of the collected data is primarily only available to the members of the research consortia but may be made available for collaborators with restrictions and only fully anonymized and pending the approval from the owners of the data

REFERENCES:
- See also: Cohort description for MADDEC consortia study plan — https://www.springerprofessional.de/en/cohort-description-for-maddec-mass-data-in-detection-and-prevent/12357640